CLINICAL TRIAL: NCT06622681
Title: Integrative Adolescence Research Programme (IARP) - iAdoRe Study
Brief Title: Integrative Adolescence Research Programme (IARP)
Acronym: IARP
Status: Recruiting | Type: Observational
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: National Institute of Education (Unknown); Nanyang Technological University (Other); Institute of High Performance Computing (IHPC), A*STAR Research Institutes (Unknown)
Responsible Party: Principal Investigator, Johan Eriksson, Executive Director, Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Other Study IDs: 2024-1200
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Executive Dysfunction; Physical Stress; Mental Health Wellness 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant of the study: Adolescents at 13- 15 years of age, currently studying in MOE-registered secondary school in Singapore and part of the DREAMS cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to understand child health during adolescence. We will examine the role of lifestyle (e.g. physical activity), growth trajectories and other environmental factors that can influence the development of phenotypes in adolescence which confer risk for later physical and mental disorders. With this study, we will develop a deeper understanding of adolescent health and well-being and their main determinants in the local Singaporean context, identify levers for early interventions to mitigate challenges to adolescent health and well-being and enhance protective factors for adolescents to do well in life, contribute to society and maximize their potential.

DETAILED DESCRIPTION:
The study aims to advance current public policy and health service practices by developing public health, clinical and commercially valuable interventions within the context of expanding commercial partnerships and building multidisciplinary translational research capacity in Singapore. In addition to the early life period (i.e., the first 1,000 days), the adolescent period has been identified as a crucial second window of opportunity to influence human development and improve life-long well-being. Adolescence is a key developmental period for body, brain and socioemotional changes. Puberty is characterised by growth spurts and sexual maturation. Concurrently, the brain undergoes maturation processes that underlie higher cognitive functions. The combination of biological changes and environmental influences affect adolescent socioemotional and behaviour patterns. There is a need to raise the human potential of adolescents who will go on to become the next generation of our adult workforce, so that they lead productive, healthy, and fulfilling lives. Yet, in many developed countries, the rates of loss of subjective well-being in young people have at least doubled in the decade prior to COVID-19 and have continued to rise since 10. In the Singapore Youth Epidemiology and Resilience Study (2020-2022), 1 in 3 youths reported experiencing mental health symptoms 11. This requires the development of a cohesive response system designed to deal with the numerous factors influencing adolescent physical and mental health. Moreover, it is essential to investigate the developmental origins of metabolic diseases and neurodevelopmental disorders, which both form a major public health burden in Singapore, from as early as the adolescence phase. A transdisciplinary approach is essential to help adolescents directly recognise their diverse concerns, challenges and experiences and better understand how to manage their health and well-being. This requires going beyond traditional psychological models of mental health to examine the influences of brain and body interaction, socio-affective, behavioural and psychological development that shape adolescents' well-being. At present, there is no comprehensive multi-disciplinary (brain-body-environment) study in the general population which examine adolescent health and well-being holistically in Asia. Findings from primarily Western countries cannot be easily extrapolated to the Singaporean/Asian setting. A new holistic programme will be essential to advance the health of Asian adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 13 to 15 years of age
2. Currently studying in MOE registered school
3. Part of the DREAMS study

Exclusion Criteria:

1. Not in MOE registered school
2. Not part of the DREAMS study

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Secondary students aged between 13 -15 years old, studying in MOE registered schools in Singapore. Part of the DREAMS study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Child health and environmental factors | 2 years
  Child's physical health and environment status
Social Science factors | 2 years
  Child's mental health status

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - A*STAR Institute for Human Development and Potential (IHDP), Singapore, Singapore
  - Singapore Institute of Clinical Sciences, Singapore

IPD SHARING:
Plan to Share IPD: No
PDPA of study participants who are minors

DOCUMENTS (2):
  • Informed Consent Form: IADORE SUB-STUDY BIOSAMPLE ICF_V1 dated 10Dec2024 (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT06622681/ICF_001.pdf
  • Informed Consent Form: IADORE SUB-STUDY BIOSAMPLE ICF (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT06622681/ICF_000.pdf